CLINICAL TRIAL: NCT02118571
Title: Schizophrenia Cognition Scale Development: Item Development and Psychometric Validation of a Novel Patient Reported Outcome (PRO) Measure for Research and Clinical Application
Brief Title: Schizophrenia Cognition Scale Development
Acronym: CIAS PRO
Status: Completed | Type: Observational
Sponsor: Carelon Research (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: P1533
Record Dates: First submitted 2014-02-25; First posted 2014-04-21 (Estimated); Last update posted 2025-02-12 (Actual); Status verified 2016-09

CONDITIONS: Schizophrenia; Cognition Disorders
MeSH Terms: conditions — Schizophrenia; Cognition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — No biospecimens collected
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this protocol is to develop items for a patient-reported outcome (PRO) measure to assess the patient's perspective and subjective experience of cognitive impairment associated with schizophrenia (CIAS).

DETAILED DESCRIPTION:
Cognitive impairment associated with schizophrenia (CIAS) has been shown to be the strongest predictor of functional impairment among people with schizophrenia because it is associated with poor response to psychosocial interventions, employment status, and social functioning. Because the subjective experience of CIAS is likely to be associated with patient burden, distress, and motivation for treatment, it is important that this experience be assessed in a reliable and valid manner and from the perspective of the patient's self report. No existing instrument to assess CIAS has been developed with patient input directly about their qualitative experience of impaired cognition during the item generation stage, in accordance with FDA guidance for patient-reported outcome (PRO) measures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with established diagnoses of schizophrenia (confirmed by the Structured Clinical Interview for DSM-IV [full version or Clinical Trial version] either performed as part of the study screening process or as documented in the medical record within 2 years prior to the study) with the following clinical features:

   * a)Clinically stable and in the residual (non-acute) phase of their illness for at least 8 weeks
   * b)Maintained on current antipsychotic and concomitant psychotropic medications for at least 6 weeks and on current dose for at least 2 weeks
   * c)Have no more than a ''moderate'' severity rating on hallucinations and delusions (e.g. Positive and Negative Syndrome Scale [PANSS] item scores < 5
   * d)Have no more than a ''moderate'' severity rating on positive formal thought disorder (e.g. Positive and Negative Syndrome Scale [PANSS] conceptual disorganization item score < 5)
   * e)Have no more than a ''moderate'' severity rating on negative symptoms (e.g., Positive and Negative Syndrome Scale-negative syndrome total score < 21)
   * f) Have no more than a minimal level of depressive symptoms (e.g. Calgary Depression Scale total score < 10); or, for eligibility for a waiting list, have a moderate level of depressive symptoms (e.g., Calgary Depression Scale total score between 10 and 15)
2. Male or female patients age 18 to 55 years
3. Exhibits reliability, physiologic capability, and an educational level sufficient to comply with all protocol procedures.
4. Able to provide informed consent

Exclusion Criteria:

1. Patient currently treated with more than two antipsychotic medications
2. Patient's cognitive impairment severity compromises the ability of the participant to participate meaningfully in a semi-structured interview, in the clinical judgment of the investigator
3. Any suicidal ideation of type 4 or 5 in the C-SSRS in the past 3 months (i.e. active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent)
4. Non-psychiatric disorders of the central nervous system (including but not limited to any kind of seizures, stroke, or traumatic brain injury)
5. Any other clinical condition that, in the opinion of the investigator, would jeopardize a patient's safety while participating in this study
6. In the 6 months prior, having met the criteria for dependence or abuse according to the DSM V in the opinion of the investigator.
7. Participation in another trial with an investigational drug or procedure within 30 days prior to screening or previous participation in any BI 409306 study
8. Unable to speak or read in English

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults with formal dx of schizo aged 18-55, stabe (non-acute phase), on stable medications
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Cognitive Impairment Associated with Schizophrenia | One time qualitative interivew within two weeks of screening
  Using qualitative interview methods, adult subjects with a diagnosis of schizophrenia will provide self reported experience of cognitive impairments associated with schizophrenia. Domains and content will be identified and explored with the subjects and used to develop the PRO measure.

SECONDARY OUTCOMES:
Assessment of Conceptual Model using Qualitative Interviews | One time qualitative interivew
  Semi structured qualitative interviews will be conducted with adult subjects with schizophrenia. The results of the interviews will be analyzed using standard methods of inductive, iterative analysis. The results will serve as the basis for generating draft items for the PRO measure.
Assess content validity and comprehension of developed PRO measure | One time qualitative interivew
  Following generation of draft PRO items, an independent series of qualitative interviews will take place in order to evaluate the draft items and ensure they accurately reflect the patient experience of cognitive impairment associated with schizophrenia.
Development and testing of a new patient reported outcome (PRO) measure | Patients will be interviewed within 2 weeks of consent
  Using qualitative interview methods, adult subjects with a diagnosis of schizophrenia will provide self reported experience of cognitive impairments associated with schizophrenia. Domains and content will be identified and explored with the subjects and used to develop the PRO measure.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond C Rosen, PhD, Principal Investigator — New England Research Institutes, Inc.
Locations (4):
- United States (4):
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Rutgers University Robert Wood Johnson Medical School, Piscataway, New Jersey
  - Richmond Behavior Associates, Staten Island, New York